CLINICAL TRIAL: NCT03557476
Title: Octacosanol Supplementation Improves Lipid Profiles and Oxidative Stress During Rapid Weight Loss and High-Intensity Exercise in Taekwondo Athletes
Brief Title: Effects of Octacosanol During Taekwondo Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kosin University (Other)
Collaborators: University of Nebraska (Other)
Responsible Party: Principal Investigator, Sang-Ho Lee, Principal Investigator, Kosin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Octacosanol
Record Dates: First submitted 2018-06-04; First posted 2018-06-15 (Actual); Results first posted 2019-08-12 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Oxidative Stress; Dyslipidemias
Keywords: Octacosanol; Taekwondo; Lipid Profiles; Oxidative Stress
MeSH Terms: conditions — Dyslipidemias | interventions — 1-octacosanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Octacosanol (Experimental): Two capsules (20-mg x 2) of 100% refined octacosanol powder from sugar cane (Swanson, Fargo ND, USA) was consumed daily by the octacosanol group for six days, one capsule 30 minutes after morning and afternoon meals.
  Interventions: Dietary Supplement: Octacosanol
- Placebo (Placebo Comparator): A placebo pill was taken twice daily in replacement of the octacosanol supplement
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Octacosanol — One capsules (20-mg) of 100% refined octacosanol powder from sugar cane (Swanson, Fargo ND, USA) was consumed twice a day
  Arms: Octacosanol
Dietary Supplement: Placebo — A placebo pill was taken twice a day in a double-blinded method at the same frequency and time as the octacosanol supplement
  Arms: Placebo

SUMMARY:
Taekwondo players undergo rapid reductions of body weight prior to their competition in order to gain a size advantage over the opponent. However, these large weight changes with concomitant high intensity exercise training induce poor lipid profiles and high levels of oxidative stress, which can be detrimental to health and sports performance. Therefore, the purpose of this study was to investigate the ability of the nutritional supplement octacosanol to combat the physiological detriments that can occur from these rapid weight changes paired with high intensity exercise training.

DETAILED DESCRIPTION:
Athletes that participate in weight division sports such as taekwondo, boxing, judo, and wrestling regularly reduce their body weight severely prior to competition in order to gain a size advantage over the opponent while simultaneously meeting their weight division requirements. In general, athletes have acute weight loss of 4-7 kg within 3-4 days of competition, while longer periods of more gradual weight loss of 15-22 kg lasting 3-4 weeks. Although this kind of extreme weight loss can induce metabolic dysfunction, it is repeatedly performed by athletes of weight division sports in order to acquire a more advantageous condition for play. Furthermore, athletes participating in matches tend to obtain excessive weights compared to their weight division during the offseason in order to lift heavier weights during training, and then rapidly lose that weight over a short period of time prior to competition, resulting in the deterioration of physiological function and possibly sports performance.

Rapid weight loss with high intensity exercise training also increases oxygen free radical production to a point that exceeds the defense mechanism of antioxidant enzymes in the body and ultimately results in damage to the cells, specifically, the lipid peroxidation of cell membranes. Not only does this decrease physiological function, but sports performance can also decrease as oxidative stress increases due to an interference in metabolic activity, a reduction in vascular function and an increase in systemic inflammation. Octacosanol, a straight-chain, high-molecular-weight, primary aliphatic alcohol minimally contained in the germinal disks of rice bran, wheat and sugar cane, may be able to prevent these deteriorations as it has been shown to provide various health benefits. In fact, previous studies reported that pre-exercise octacosanol intake contributed to enhanced muscular strength, muscular endurance and oxygen transport ability. Additionally, octacosanol supplementation has been shown to improve cardiovascular endurance and heart function in patients with peripheral artery disease, improve levels of low-density and high-density lipoprotein-cholesterol in patients with hypercholesterolemia, and increase glycogen accumulation in mice9. However, the potential beneficial effects of octacosanol intake for reducing free radical production and preventing detrimental physiological function from excessive weight loss with high intensity exercise has not been examined. Thus, the purpose of this study was to investigate the effects of octacosanol supplementation during acute weight loss with high-intensity exercise training on lipid profiles and markers of oxidative stress in taekwondo players.

ELIGIBILITY:
Inclusion Criteria:

* at least 3 years of experience in national taekwondo competitions
* abstain from caffeinated drinks, alcohol, and antioxidant supplements during the whole period of the study

Exclusion Criteria:

* no history of chronic use of antioxidants, chronic aspirin, and nonsteroidal anti-inflammatory drugs (NSAIDs)
* No cardiovascular, neurological, metabolic or renal diseases
* no musculoskeletal injuries

Ages: 17 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Song Park, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska at Omaha, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Octacosanol | Placebo
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Octacosanol | Placebo | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 18 (1) | 18 (1) | 18 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 13 | 13 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 13 | 26
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 13 | 13 | 26
Height [Mean (Standard Deviation); unit: cm] | 174.7 (1.4) | 173.9 (6.3) | 174.3 (3.9)
Weight [Mean (Standard Deviation); unit: kg] | 66.9 (6.7) | 66.7 (5.7) | 66.8 (6.2)
Body fat [Mean (Standard Deviation); unit: percentage of body fat] | 8 (2) | 8 (2) | 8 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Triglycerides
Description: Plasma triglyceride levels
Time Frame: 6 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Octacosanol | Placebo
Number analyzed (Participants) | 13 | 13
mg/dL | 34.9 (7.8) | 110 (8.1)

2. Primary Outcome: Total Cholesterol
Description: Plasma total cholesterol levels
Time Frame: 6 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Octacosanol | Placebo
Number analyzed (Participants) | 13 | 13
mg/dL | 164 (12.8) | 173.5 (16.1)

3. Primary Outcome: High-density Lipoprotein
Description: Plasma levels of high-density lipoprotein
Time Frame: 6 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Octacosanol | Placebo
Number analyzed (Participants) | 13 | 13
mg/dL | 71 (4.4) | 49.2 (2.6)

4. Primary Outcome: Low-density Lipoprotein
Description: Plasma levels of low-density lipoprotein
Time Frame: 6 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Octacosanol | Placebo
Number analyzed (Participants) | 13 | 13
mg/dL | 92.6 (8.1) | 114.9 (10.8)

5. Secondary Outcome: Malondialdehyde
Description: Plasma levels of malondialdehyde
Time Frame: 6 days
Measure: Mean (Standard Deviation); unit: mmol/mL
Arm/Group | Octacosanol | Placebo
Number analyzed (Participants) | 13 | 13
mmol/mL | 0.25 (0.1) | 0.93 (0.12)

6. Secondary Outcome: Superoxide Dismutase
Description: Plasma levels of superoxide dismutase
Time Frame: 6 days
Measure: Mean (Standard Deviation); unit: U/gHb
Arm/Group | Octacosanol | Placebo
Number analyzed (Participants) | 13 | 13
U/gHb | 1450 (138.9) | 1010 (150.1)

7. Secondary Outcome: Glutathione Peroxidase
Description: Plasma levels of glutathione peroxidase
Time Frame: 6 days
Measure: Mean (Standard Deviation); unit: U/gHb
Arm/Group | Octacosanol | Placebo
Number analyzed (Participants) | 13 | 13
U/gHb | 66.9 (10.8) | 47.1 (9.7)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Octacosanol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/76/NCT03557476/Prot_SAP_000.pdf